CLINICAL TRIAL: NCT03928301
Title: Efficacy of Wholetones® 2Sleep Music on Health and Sleep Behaviors of Healthy Adults With Insomnia Symptoms: A Single Blind Randomized Controlled Crossover Trial
Brief Title: Efficacy of Wholetones® 2Sleep Music on Health and Sleep Behaviors of Healthy Adults With Insomnia Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacksonville University (Other)
Responsible Party: Principal Investigator, Dr. Heather Hausenblaus, Lead Investigator, Jacksonville University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 363968-1
Record Dates: First submitted 2019-04-12; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Insomnia; Sleeplessness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wholetones Intervention (Active Comparator): Wholetones music to help participants sleep. Data collected after listening to the Wholetones music was compared to that collected both at Baseline, and after listening to the other music condition (i.e. Classical music).
  Wholetones® 2Sleep is music that is designed to lull the listener into a deep, delta sleep, using frequency-enhanced music and precise tempos. Wholetones® differs from other musical genres in that it employs a proprietary method of tuning and layering the music with a unique frequency underlayment.
  Interventions: Behavioral: Wholetones Music
- Classical Intervention (Active Comparator): Classical music was the additional music condition used to compare to both Baseline data and Wholetones data.
  The classical music was selected based on the Mayo Clinic and NIH music recommendations for better sleep. More specifically, the classical music consisted of the following six pieces: Beethoven (i.e., Moonlight Sonata, first movement), Marconi Union (i.e., Weightless), Chopin (i.e., Nocturne No.2, Op.9), Ravel (i.e., Piano Concerto in G major, 2nd movement), and J.S. Bach (i.e., Prelude No.1).
  Interventions: Behavioral: Classical Music

INTERVENTIONS:
Behavioral: Wholetones Music — Participants listened to the Wholetones music for 10 nights consecutively. Participants began playing the music 30 minutes before going to bed and were asked to allow it to play continuously throughout the night.
  Arms: Wholetones Intervention
Behavioral: Classical Music — Participants listened to the classical music for 10 nights consecutively. Participants began playing the music 30 minutes before going to bed and were asked to allow it to play continuously throughout the night.
  Arms: Classical Intervention

SUMMARY:
(b) The investigators propose to conduct a four-week randomized controlled crossover trial on healthy adults with occasional sleeplessness to examine the efficacy of Wholetones music on their health-related quality of life, sleep quality and quantity, anxiety/stress levels, mood, and EMFIT sleep tracker data. Baseline sleep data will be obtained for the first week of the study. Using a crossover design, each participant will then be randomized for 10 days to each of the following two conditions: (1) Wholetones music and (2) classical music. The participants will be instructed to listed to the music for 30 minutes prior to sleep each night. The self-report assessments will be taken at Day 0 (baseline), Day 7, Day 17, Day 21, and Day 31. The participants will also complete a sleep daily survey and use the EMFIT tracker nightly. It is hypothesized that the music conditions will result in improved sleep behaviors and self-report health outcomes compared to the classical music condition. It is also hypothesized that a dose-response will be evidenced with stronger effects found for Wholetones music compared to the classical music.

DETAILED DESCRIPTION:
To determine if the Wholetones® or classical music was successful at alleviating symptoms of insomnia or sleeplessness when compared to not listening to any music, self-report data from large surveys was collected both at baseline, and during the interventions at day 17 (after the first music condition), and at day 31 (after the second music condition. Participants also completed daily diaries which was comprised of 6 questions that assessed their music adherence, sleep quality, and music likeability. These were completed daily from baseline through to the end of the study.

Objective data was also collected during baseline period of 1-week, throughout both of the interventions (10 nights each for a total of 20 nights) and the washout period (4 nights) using the EMFIT tracker. This device relies on ballistocardiography, was used to objectively assess nighttime sleep in the natural environment. This sleep tracker is automatic, autonomous, and is installed under the mattress.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia Index score indicating occasional sleeplessness

Exclusion Criteria:

* BMI over 34
* smokers
* heart conditions
* sleep apnea

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Change In Pittsburgh Sleep Quality Index Scores from Baseline to those at Days 17 & 31 | Day 0, Day 17 (following 10 days of one music condition), Day 31 (following 10 days of second music condition)
  Self report data used to determine how well participants perceived their sleep quality at Day 0 (baseline), Day 17 (after first music condition Wholetones or classical), and Day 31 (after alternate music condition). This survey consists of 9 total items (some items have sub questions i.e. item 4 which has parts A and B). Scores are calculated as per survey instructions. Any scores of 5 or above indicate poor perceived sleep quality.
Change In Profile of Mood States (POMS) Scores from Baseline to Days 17 & 31 | Day 0, Day 17 (following 10 days of one music condition), Day 31 (following 10 days of second music condition)
  Self report data used to determine the perceived mood of participants at Day 0 (baseline), Day 17 (after first music condition Wholetones or classical), and Day 31 (after alternate music condition). This questionnaire has 65 total items and responses are calculated by scoring question responses on a Likert scale fro 0-4, where 0= not at all and 4= extremely. Total numeric scores are determined for the 6 sub scales represented in the survey (i.e. depression, anger, vigor, confusion, tension, and anger) based on which category the item represents. These sub scale scores are then tallied to determine and overall mood score, where higher scores indicate higher levels of depression, anger, tension, confusion, and fatigue. Being that vigor is a positive indicator for mood, these items are reverse scored before being tallied.
Change in State Trait Anxiety Inventory Scores from Baseline to Days 17 & 31 | Day 0, Day 17 (following 10 days of one music condition), Day 31 (following 10 days of second music condition)
  Self report data used to determine the perceived anxiety levels of participants at Day 0 (baseline), Day 17 (after first music condition Wholetones or classical), and Day 31 (after alternate music condition). This survey has 20 total items, and responses are scored on a Likert scale of 1-4 where 1=almost never and 4=almost always. Any items that are positive are reverse scored before totaling all 20 items. Higher scores indicate higher levels of perceived anxiety.
Change In Perceived Stress Scale Scores at Baseline from Days 17 & 31 | Day 0, Day 17 (following 10 days of one music condition), Day 31 (following 10 days of second music condition)
  Self report data used to determine the perceived stress levels of participants at Day 0 (baseline), Day 17 (after first music condition Wholetones or classical), and Day 31 (after alternate music condition). This survey has 10 total items, and responses are scored on a Likert scale from 0-4 where 0=Never and 4=Very often. Any items that are positive are reverse scored before totaling all 10 items. Higher scores indicate higher levels of perceived stress.
Change In Flinder's Fatigue Scale Scores from Baseline to Days 17 & 31 | Day 0, Day 17 (following 10 days of one music condition), Day 31 (following 10 days of second music condition)
  Self report data used to determine the perceived fatigue levels of participants at Day 0 (baseline), Day 17 (after first music condition Wholetones or classical), and Day 31 (after alternate music condition). This survey has 7 total items, and 6 out of the 7 items are scored on a 5-point Likert scale of 0 (Not at all) to 4 (Extremely). The 7th item asks participants during which times of day they typically experience the most fatigue (out of 7 possible options), each time that indicate is counted as a "1" and all times selected are added to determine a score for that item. All 7 items are then tallied to determine a final score, where higher scores indicate higher levels of perceived fatigue.
Change In Productivity Scores from Baseline to Days 17 & 31 | Day 0, Day 17 (following 10 days of one music condition), Day 31 (following 10 days of second music condition)
  Self report data used to determine the perceived productivity levels of participants at Day 0 (baseline), Day 17 (after first music condition Wholetones or classical), and Day 31 (after alternate music condition). This was determined using 1 item from a Life Satisfaction survey. It was scored using a Likert scale where 1 represented "Very Unproductive" and 4 "Very Productivity". Higher scores indicate higher levels of perceived productivity.
EMFIT Sleep Tracker data | This data was collected for the 1-month duration of the study (7 days of baseline, 20 days of intervention, 4 days of washout).
  EMFIT sleep tracker reports served as the objective sleep data for the study. Sleep data was collected during the night while participants slept in their own beds. The EMFIT tracker has a sensor strip that goes underneath the participant's mattress, which is connected to a small senor device that plugs into the wall near the bed, and which connects the the participant's WiFi in order to transmit sleep data. This device was used to measure heart rate, breathing rate, movement activity every 4 seconds, sleep staging every 30 seconds, and heart rate variability every 3 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Jacksonville University, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ancoli-Israel S, Roth T. Characteristics of insomnia in the United States: results of the 1991 National Sleep Foundation Survey. I. Sleep. 1999 May 1;22 Suppl 2:S347-53. PMID 10394606
- [Background] Buysse DJ, Ancoli-Israel S, Edinger JD, Lichstein KL, Morin CM. Recommendations for a standard research assessment of insomnia. Sleep. 2006 Sep;29(9):1155-73. doi: 10.1093/sleep/29.9.1155. PMID 17040003
- [Background] Chang ET, Lai HL, Chen PW, Hsieh YM, Lee LH. The effects of music on the sleep quality of adults with chronic insomnia using evidence from polysomnographic and self-reported analysis: a randomized control trial. Int J Nurs Stud. 2012 Aug;49(8):921-30. doi: 10.1016/j.ijnurstu.2012.02.019. Epub 2012 Apr 10. PMID 22494532
- [Background] Jespersen KV, Otto M, Kringelbach M, Van Someren E, Vuust P. A randomized controlled trial of bedtime music for insomnia disorder. J Sleep Res. 2019 Aug;28(4):e12817. doi: 10.1111/jsr.12817. Epub 2019 Jan 24. PMID 30676671
- [Background] de Niet G, Tiemens B, Lendemeijer B, Hutschemaekers G. Music-assisted relaxation to improve sleep quality: meta-analysis. J Adv Nurs. 2009 Jul;65(7):1356-64. doi: 10.1111/j.1365-2648.2009.04982.x. Epub 2009 Apr 28. PMID 19456998
- [Background] Feng F, Zhang Y, Hou J, Cai J, Jiang Q, Li X, Zhao Q, Li BA. Can music improve sleep quality in adults with primary insomnia? A systematic review and network meta-analysis. Int J Nurs Stud. 2018 Jan;77:189-196. doi: 10.1016/j.ijnurstu.2017.10.011. Epub 2017 Oct 23. PMID 29100201
- [Background] Harmat L, Takacs J, Bodizs R. Music improves sleep quality in students. J Adv Nurs. 2008 May;62(3):327-35. doi: 10.1111/j.1365-2648.2008.04602.x. PMID 18426457
- [Background] Huang CY, Chang ET, Lai HL. Comparing the effects of music and exercise with music for older adults with insomnia. Appl Nurs Res. 2016 Nov;32:104-110. doi: 10.1016/j.apnr.2016.06.009. Epub 2016 Jun 23. PMID 27969011
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Trahan T, Durrant SJ, Mullensiefen D, Williamson VJ. The music that helps people sleep and the reasons they believe it works: A mixed methods analysis of online survey reports. PLoS One. 2018 Nov 14;13(11):e0206531. doi: 10.1371/journal.pone.0206531. eCollection 2018. PMID 30427881
- [Result] Jespersen KV, Koenig J, Jennum P, Vuust P. Music for insomnia in adults. Cochrane Database Syst Rev. 2015 Aug 13;2015(8):CD010459. doi: 10.1002/14651858.CD010459.pub2. PMID 26270746